CLINICAL TRIAL: NCT00048737
Title: Safety and Efficacy of 90Y Zevalin in Nonmyeloablative Transplantation for Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-233
Record Dates: First submitted 2002-11-06; First posted 2002-11-08 (Estimated); Results first posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma; Leukemia
Keywords: Leukemia; Lymphoma; Lymphoid Malignancy; Cyclophosphamide; Cytoxan; Neosar; Fludarabine; Fludarabine Phosphate; Fludara; Rituximab; Rituxan; Zevalin; Indium Zevalin; 90Y Zevalin; CD-20-positive; B-cell Lymphoma; CD-20-positive B-cell Lymphoma; NHL; CLL; Chronic Lymphocytic Leukemia; Allogeneic Stem Cell Transplantation; ASCT
MeSH Terms: conditions — Lymphoma; Leukemia; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 90Y Zevalin in ASCT (Experimental): Allogeneic Stem Cell (AST) Transplantation with 90Y Zevalin/Cyclophosphamide/Fludarabine as a preparative regimen.
  Interventions: Drug: Zevalin Radioimmunotherapy; Drug: Rituximab; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Allogeneic Stem Cell Transplantation

INTERVENTIONS:
Drug: Zevalin Radioimmunotherapy — Escalating single dose of 90Y Zevalin 0.2-0.3-0.4 mCi/kg
  Other Names: 90Y Zevalin
Drug: Rituximab — 250 mg/m^2 on day 1 and day 8
  Other Names: Rituxan
Drug: Fludarabine — 30 mg/m^2/day for 3 days
  Other Names: Fludarabine phosphate; Fludara
Drug: Cyclophosphamide — 750 mg/m^2/day for 3 days, given on the same days as fludarabine, at 4-hour intervals
  Other Names: Cytoxan; Neosar
Procedure: Allogeneic Stem Cell Transplantation — Allogeneic stem cell transplantation 2 days after chemotherapy
  Other Names: ASCT

SUMMARY:
The goal of this clinical research study is to see if low intensity chemotherapy given together with the new drug 90Y Zevalin, followed by a transplant of blood or marrow stem cells from a donor can increase the length of remission in patients with leukemia and lymphoma. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Rituxan is an antibody made from human and mouse protein. It reacts with a certain antigen on lymphoma cells and causes the body's immune system to destroy the lymphoma cells. 90Y Zevalin and 111In Zevalin are murine-based antibodies combined with a radioactive agent that can also destroy lymphoma cells. Unlike Rituxan, 90Y Zevalin cannot be traced by regular scanning and requires indium to determine its distribution through the body.

Before treatment starts, patients will have a physical exam, including blood tests and urine tests. Women who are able to have children must have a negative blood pregnancy test. Bone marrow samples will be taken. For bone marrow sampling, a large needle is placed in the hipbone after it has been numbed. The bone marrow is then withdrawn through the needle. Patients will have a chest x-ray, computed tomography (CT) scans, an EKG, and tests of lung function.

Blood tests, urine tests, bone marrow sampling, and x-rays will be done as needed to track the effects of the transplant. Patients will have transfusions of blood and platelets as needed. Blood tests will be done daily while patients are in the hospital.

Patients in this study will receive an unlabeled antibody form of Y2B8 called rituxan by vein followed by a dose of 111In Zevalin by vein. 111In Zevalin includes the radioactive agent indium, which shows up when patients have x-rays or scans. The scans can show where and how fast the drug travels in the body and how long the drug stays in the body. Doctors need to be able to see how much of the drug goes to the tumor and how much goes to normal organs to see if it is safe to give 90Y Zevalin on an outpatient basis. A scan will be taken 48 to 72 hours after 111In Zevalin is given.

If the radiation in the 111In Zevalin is not a threat to normal organs and bone marrow, patients may receive 90Y Zevalin. Seven days after the 111In Zevalin injection, patients will receive a second dose of rituxan followed by a dose of 90Y Zevalin.

Patients will also receive fludarabine and cyclophosphamide daily for 3 days. All of the chemotherapy drugs will be given through a catheter (plastic tube) that extends into the large chest vein. The catheter will be left in place throughout treatment. When chemotherapy is finished, blood stem cells from a donor will be given through the catheter. Granulocyte colony-stimulating factor (G-CSF or GCSF), a hormone that helps the production of blood cells, will be injected under the skin once a day until the neutrophil counts recover in the blood. Patients will receive methotrexate for 3 days post transplant and tacrolimus for 6 months or more to prevent graft versus host disease.

All patients will have complete checkups, including blood and urine tests 2 or 3 times during the first 12 weeks of the study. Tumors will be measured by CT or MRI and gallium scans. Patients will be asked to fill out a survey about quality of life issues (maintaining normal routine, family life, social life, pain). It takes about half an hour to fill out the survey. A bone marrow sample may be taken. A test of heart function will be done. Checkups and tests will be done every 3 months for 1 year and then every 6 months for 4 more years.

Treatment will be given in the hospital at M. D. Anderson. Patients will need to stay in the hospital for about 3 to 4 weeks. Patients must stay in the Houston area for about 100 days after the transplant. After that, patients will need to return to Houston from time to time for blood tests, urine tests, and other exams.

This is an investigational study. 90Y-Zevalin is approved by the FDA for relapsed and refractory lymphoma. Its use in this trial, however, is investigational. About 70 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in relapse or considered at high risk for relapse or refractory CD-20-positive B-cell NHL or CLL. Patients considered for high risk of relapse are patients who do not achieve complete response (CR) with frontline chemotherapy, CLL is Richter's and CLL with high risk chromosomal abnormalities.
2. Measurable disease.
3. Age 18-70 years, expected survival >/= 3 months, performance status 0 to 2.
4. Availability of a matched related donor.
5. </+ 50% bone marrow involvement.
6. CLL with </+ 10,000 circulating lymphocytes.
7. Availability of a matched related or unrelated donor.

Exclusion Criteria:

1. Prior myeloablative therapies or radioimmunotherapy.
2. Prior external beam radiation therapy to >25% of active bone marrow.
3. Prior therapy with 90Y Zevalin or Campath.
4. CNS lymphoma, HIV, HTLV-1 positivity, some creatinine >1.6 mg/dl or serum bilirubin >1.5 mg/dl.
5. Pregnancy or lactation.
6. Symptomatic pulmonary or cardiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Khouri IF, Saliba RM, Erwin WD, Samuels BI, Korbling M, Medeiros LJ, Valverde R, Alousi AM, Anderlini P, Bashir Q, Ciurea S, Gulbis AM, de Lima M, Hosing C, Kebriaei P, Popat UR, Fowler N, Neelapu SS, Samaniego F, Champlin RE, Macapinlac HA. Nonmyeloablative allogeneic transplantation with or without 90yttrium ibritumomab tiuxetan is potentially curative for relapsed follicular lymphoma: 12-year results. Blood. 2012 Jun 28;119(26):6373-8. doi: 10.1182/blood-2012-03-417808. Epub 2012 May 14. PMID 22586182
- See also: The University of Texas M.D.Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 30, 2002 to September 21, 2010. All participants were recruited at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- 90Y Zevalin in ASCT: Allogeneic Stem Cell (AST) Transplantation with 90Y Zevalin/Cyclophosphamide/Fludarabine as a preparative regimen.
  Rituximab : 250 mg/m^2 on day 1 and day 8
  Allogeneic Stem Cell Transplantation : Allogeneic stem cell transplantation 2 days after chemotherapy
  Cyclophosphamide : 750 mg/m^2/day x 3, given on the same days as fludarabine, at 4-hour intervals
  Zevalin Radioimmunotherapy : Escalating single dose of 90Y Zevalin 0.2-0.3-0.4 mCi/kg
  Fludarabine : 30 mg/m^2/day x 3
Period: Overall Study
Arm/Group | 90Y Zevalin in ASCT
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 90Y Zevalin in ASCT
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Failure
Description: Graft failure is defined as either lack of hematologic recovery or lack of or loss of detectable donor cells.
Time Frame: 100 days
Measure: Number; unit: participants
Groups:
- 90Y Zevalin in ASCT: Allogeneic Stem Cell (AST) Transplantation with 90Y Zevalin/Cyclophosphamide/Fludarabine as a preparative regimen.
  Rituximab: 250 mg/m^2 on day 1 and day 8
  Allogeneic Stem Cell Transplantation : Allogeneic stem cell transplantation 2 days after chemotherapy
  Cyclophosphamide : 750 mg/m^2/day x 3, given on the same days as fludarabine, at 4-hour intervals
  Zevalin Radioimmunotherapy : Escalating single dose of 90Y Zevalin 0.2-0.3-0.4 mCi/kg
  Fludarabine : 30 mg/m^2/day x 3
Arm/Group | 90Y Zevalin in ASCT
Number analyzed (Participants) | 70
participants | 1

ADVERSE EVENTS:
Time Frame: 9 Years and 1 Month
Arm/Group | 90Y Zevalin in ASCT
Serious Adverse Events (participants affected / at risk) | 7/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 90Y Zevalin in ASCT (N=70)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — # of participants affected-1
Thrombosis (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
C-Diff Colitis (Gastrointestinal disorders) | 1 (1)
Viral Hepatitis B reactivation (Infections and infestations) | 1 (1)
secondary malignancy- Melanoma (Skin and subcutaneous tissue disorders) | 1 (1)
Right Inguinal hernia (General disorders) | 1 (1)
Prolonged Hospitalization, Generalized Weakness/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death due to G.I. GVHD (Gastrointestinal disorders) | 1 (1)
Secondary Malignancy-Early Nodular Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Death Due to Chronic Liver/G.I GVHD (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 90Y Zevalin in ASCT (N=70)
Neuoropathy (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 61 (61)
Diarrhea (Gastrointestinal disorders) | 28 (28)
Mucositis (Gastrointestinal disorders) | 22 (22)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 12 (12)
Elevated ALT (Hepatobiliary disorders) | 16 (16)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 10 (10)
Increased Bilirubin (Hepatobiliary disorders) | 7 (7)
Increased LDH (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 37 (88)
Hypertension (Cardiac disorders) | 10 (10)
Edema (Cardiac disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 1 (1)
Low Ejection Fraction (Cardiac disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 9 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 12 (12)
Dizziness (Nervous system disorders) | 1 (1)
Altered Mood (Nervous system disorders) | 3 (3)
Insomnia (Nervous system disorders) | 3 (3)
Pain (Nervous system disorders) | 5 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 32 (32)
Skin Dryness (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 21 (21)
Fatigue (General disorders) | 6 (6)
Rigors (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Altered Mood-Agitation (Nervous system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Fasciitis (Skin and subcutaneous tissue disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No